CLINICAL TRIAL: NCT06198816
Title: Inflow Improve for Deep Vein ThrombOsis with Ultrasound AcceLerated ThrombOlysis and Venoplasty: a Monocentric, Observational and Prospective Study.
Brief Title: Inflow Improve for Deep Vein ThrombOsis with Ultrasound AcceLerated ThrombOlysis and Venoplasty
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Baccellieri Domenico, Principal Investigator, IRCCS San Raffaele
Other Study IDs: IDOLO Study
Record Dates: First submitted 2023-12-28; First posted 2024-01-10 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Post-Thrombotic Syndrome of Both Legs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- DVT patients
  Interventions: Other: ultrasound accelerated thrombolysis and venoplasty

INTERVENTIONS:
Other: ultrasound accelerated thrombolysis and venoplasty — IDOLO Study investigate clinical efficacy on ultrasound accelerated thrombolysis and venoplasty in patients with post-thrombotic syndrome secondary to chronical femoro-popliteal vein occlusion for previous deep vein Thrombosis (DVT).

SUMMARY:
Aim of the IDOLO study is to investigate clinical efficacy on ultrasound accelerated thrombolysis and venoplasty in patients with post-thrombotic syndrome secondary to chronical femoro-popliteal vein occlusion for previous deep vein Thrombosis (DVT).

At San Raffaele Hospital (Vascular Surgery Department) will be enrolled 50 patients with lower extremity deep vein thrombosis (who have failed conservative treatment) objectively diagnosed with imaging ≥ 6 months; prior persistent deep vein Thrombosis (DVT) at enrollment evaluation and moderate-severe post-thrombotic syndrome at time of procedure

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted in Vascular Surgery Unit, San Raffaele Hospital, Milan
* Patients able to sign specific informed consent for the study.
* Proximal deep vein Thrombosis (iliac vein, common femoral vein, deep femoral vein, and femoral vein) that was objectively diagnosed with duplex imaging and/or venography ≥ 6 months prior to study screening.
* Persistent chronic deep vein Thrombosis causing restrictive flow, as confirmed by imaging, within 60 days prior to the study procedure.
* Failed a minimum of 3 consecutive months of conservative treatment (therapeutic anticoagulation and compression stockings).
* Villalta score ≥8 for the affected limb within 30 days prior to the study procedure

Exclusion Criteria:

* Treated with mechanical thrombectomy within 2 weeks of the study thrombolysis procedure.
* Treated with thrombolysis drugs within 48 hours of the study thrombolytic procedure.
* Life expectancy less than (<) 1 year.
* Body Mass Index (BMI) greater than (>) 40 kilograms/square meter (kg/m^2) or per Investigator's discretion participant is able tolerate the procedure and be compliant with post-procedure increased physical activity.
* No flow in popliteal vein on duplex imaging
* Thrombus extending ≥ 3 centimeters (cm) into the inferior vena cava (IVC). If central venous occlusion, consider computed tomography (CT) or magnetic resonance venography (MRV). For participants with bilateral DVT, it is recommended that central imaging be performed prior to treatment to evaluate the status of the IVC.
* Active bleeding, recent (<3 months) gastrointestinal (GI) bleeding, active peptic ulcer, severe liver dysfunction, and bleeding diathesis.
* Recent (<3 months) internal eye surgery or hemorrhagic retinopathy; recent (<10 days) major surgery, cataract surgery, trauma, cardiopulmonary resuscitation (CPR), obstetrical delivery, or other invasive procedure.
* History of stroke or intracranial/intraspinal bleed, tumor, vascular malformation, or aneurysm.
* Active cancer (metastatic, progressive, or treated within the last 6 months). Participants with non-melanoma primary skin cancers are eligible to participate in the study.
* Hemoglobin <9.0 milligrams/deciliter (mg/dL) within 24 hours prior to the procedure
* International normalized ratio (INR) ≥1.5 nanograms/deciliter (ng/dL) within 24 hours prior to the procedure.
* Platelet count <100,000 cells/cubic millimeter (cells/mm^3) or >700,000 cells/mm^3 within 24 hours prior to the procedure.
* Creatinine outside the normal range for the treating institution and considered clinically significant by the Investigator.
* Uncontrolled hypertension, defined as systolic >175 millimeters of mercury (mmHg) and a diastolic >110 mmHg.
* Use of clopidogrel, ticlopidine, or other thienopyridine antiplatelet drug within 7 days of the study procedure.
* In the judgment of the clinician, the participant is at high risk for catastrophic bleeding.
* Impossibility or refusal to give informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: At San Raffaele Hospital (Vascular Surgery Department) will be enrolled 50 patients with lower extremity deep vein thrombosis (who have failed conservative treatment) objectively diagnosed with imaging ≥ 6 months; prior persistent DVT at enrollment evaluation and moderate-severe post-thrombotic syndrome at time of procedure.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Clinical Severity Scores | up to 12 months
  Improvement of Clinical efficacy will be evaluated using the Villalta score
Major Bleeding | 72 hours
  Freedom from Fatal bleeding, Symptomatic bleeding in a critical area or organ,Bleeding causing a fall in hemoglobin level of 20gL

CONTACTS AND LOCATIONS:
Locations (1):
- San Raffaele Hospital, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garcia MJ, Sterling KM, Kahn SR, Comerota AJ, Jaff MR, Ouriel K, Weinberg I; ACCESS PTS Investigators. Ultrasound-Accelerated Thrombolysis and Venoplasty for the Treatment of the Postthrombotic Syndrome: Results of the ACCESS PTS Study. J Am Heart Assoc. 2020 Feb 4;9(3):e013398. doi: 10.1161/JAHA.119.013398. Epub 2020 Jan 25. PMID 31983322
- [Background] Grommes J, Strijkers R, Greiner A, Mahnken AH, Wittens CH. Safety and feasibility of ultrasound-accelerated catheter-directed thrombolysis in deep vein thrombosis. Eur J Vasc Endovasc Surg. 2011 Apr;41(4):526-32. doi: 10.1016/j.ejvs.2010.11.035. Epub 2011 Jan 21. PMID 21256773
- [Background] Shi Y, Shi W, Chen L, Gu J. A systematic review of ultrasound-accelerated catheter-directed thrombolysis in the treatment of deep vein thrombosis. J Thromb Thrombolysis. 2018 Apr;45(3):440-451. doi: 10.1007/s11239-018-1629-y. PMID 29417407
- [Background] Dumantepe M, Tarhan IA, Ozler A. Treatment of chronic deep vein thrombosis using ultrasound accelerated catheter-directed thrombolysis. Eur J Vasc Endovasc Surg. 2013 Sep;46(3):366-71. doi: 10.1016/j.ejvs.2013.05.019. Epub 2013 Jun 25. PMID 23806796